CLINICAL TRIAL: NCT06285578
Title: Effects of Probiotic With HIIT on Cardiorespiratory Endurance and Metabolism in Middle-Aged Obese Women
Brief Title: Effects of Probiotic and HIIT in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taipei (Other)
Responsible Party: Principal Investigator, Chien-Wen Hou, Principle investigator, University of Taipei
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MOST 107-2410-H-277-003
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cardiorespiratory Fitness; Metabolism; Anthropometry

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo control (C) (Placebo Comparator): The subjects do not perform HIIT training, but consume one placebo packet every day on a fasting status for 8 weeks.
  Interventions: Dietary Supplement: Placebo supplementation
- Probiotics supplementation (P) (Experimental): Each participant consume one probiotic packet every day on a fasting status for 8 weeks.
  Interventions: Dietary Supplement: Probiotics supplementation
- HIIT intervention (H) (Experimental): HIIT training for 3 sessions per week and consume one placebo packet every day on a fasting status for 8 weeks.
  Interventions: Behavioral: HIIT training; Dietary Supplement: Placebo supplementation
- HIIT with probiotics intervention (HP) (Experimental): Conduct HIIT training 3 sessions per week for 8 weeks and consume one probiotic packet every day on a fasting status for 8 weeks.
  Interventions: Dietary Supplement: Probiotics supplementation; Behavioral: HIIT training

INTERVENTIONS:
Dietary Supplement: Probiotics supplementation — Probiotics, Lactiplantibacillus plantarum TWK10, are packaged in powder form. Each participant consume one packet every day on a fasting status for 8 weeks.
  Arms: HIIT with probiotics intervention (HP); Probiotics supplementation (P)
Behavioral: HIIT training — HIIT training is conduct at the intensity of 85-90% VO2max for 2 minutes with 1-minute inactive resting interval, repeating for 7 times. 3 sessions per week for 8 weeks.
  Arms: HIIT intervention (H); HIIT with probiotics intervention (HP)
Dietary Supplement: Placebo supplementation — Yeast powder replaces probiotics in each packet. Each participant consume one packet every day on a fasting status for 8 weeks.
  Arms: HIIT intervention (H); Placebo control (C)

SUMMARY:
The aim of this study is to investigate whether there are the additive effects when implementing both high-intensity interval training (HIIT) and probiotics simultaneously on improving cardiorespiratory endurance and metabolism in middle-aged women.

DETAILED DESCRIPTION:
High-intensity interval training (HIIT) is a time-efficiency exercise mode that has been shown to reduce body fat, fasting blood insulin levels, arterial stiffness, and aerobic capacity, helping to prevent and improve chronic diseases. Probiotics, on the other hand, have been found to have similar effects, including improving insulin sensitivity and endurance exercise performance, as well as reducing body fat. However, the additive effects of HIIT combined with probiotic supplements are unclear. In addition, on average, the life expectancy of women is longer than that of men. Middle-aged women are at high-risk for obesity and metabolic-related problems that threaten their long-term health. Therefore, whether the combination of HIIT and probiotics can be utilized to enhance the wellness of middle-aged women is the objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age between 35-55 years old
* Total body fat percentage greater than 30%

Exclusion Criteria:

* Male
* Participants who were taking probiotics supplementation or antibiotics
* Percentage of total body fat less than 30%

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Height | 8 weeks
  Height in centimeters
Body weight | 8 weeks
  Weight in kilograms
Body mass index (BMI) | 8 weeks
  Calculated by: weight (kg)/ height (m^2)
Body fat percentage | 8 weeks
  Body fat percentage (%) is measured with Dual-energy X-ray absorptiometry (DEXA)
Waist circumference | 8 weeks
  Waist circumference in centimeters
Hip circumference | 8 weeks
  Hip circumference in centimeters
Maximum oxygen uptake (VO2max) | 8 weeks
  VO2max in ml/min/kg
Time to exhaustion (TTE) | 8 weeks
  TTE in seconds
Running economy (RE) | 8 weeks
  RE in ml/kg/km
Fasting blood glucose (FBG) | 8 weeks
  FBG in mg/dL
Total cholesterol (TC) | 8 weeks
  TC in mg/dL
Triglyceride (TG) | 8 weeks
  TG in mg/dL
High-density lipoprotein cholesterol (HDL-C) | 8 weeks
  HDL-C in mg/dL
Low-density lipoprotein cholesterol (LDL-C) | 8 weeks
  LDL-C in mg/dL

SECONDARY OUTCOMES:
Muscle mass | 8 weeks
  Muscle mass in kilograms is measured with DEXA
Fat mass | 8 weeks
  Fat mass in kilograms is measured with DEXA
Bone mineral density (BMD) | 8 weeks
  BMD in g/cm^2 is measured with DEXA
Caloric intake | 8 weeks
  Caloric intake in kcal/day

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Wen Hou, Ph.D., Study Director — University of Taipei
Locations (1):
- University of Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Chen YC, Wang HY, Ogita F, Hung CH, Kuo CH, Wang JP, Wang CM, Hou CW, Wang TY. Effects of probiotic supplementation with high-intensity interval training on cardiorespiratory endurance and metabolism in Middle-Aged Obese Women. J Int Soc Sports Nutr. 2024 Dec;21(1):2425609. doi: 10.1080/15502783.2024.2425609. Epub 2024 Dec 1. PMID 39618097